CLINICAL TRIAL: NCT02501954
Title: Randomized Phase III Trial of Cisplatin and Tumor Volume Directed Irradiation Followed by Carboplatin and Paclitaxel Vs. Sandwich Therapy of Carboplatin and Paclitaxel Followed by Tumor Volume Directed Irradiation Then Further Carboplatin and Paclitaxel
Brief Title: Trial of Cisplatin Plus Radiation Followed by Carbo and Taxol Vs. Sandwich Therapy of Carbo and Taxol Followed Radiation Then Further Carbo and Taxol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Women's Cancer Care Associates, LLC (Other)
Responsible Party: Principal Investigator, Joyce N. Barlin, MD, Principal Investigator, Women's Cancer Care Associates, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-07
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Stage IIIA Uterine Corpus Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC Uterine Corpus Cancer; Stage IVA Uterine Corpus Cancer
MeSH Terms: interventions — Cisplatin; Carboplatin; Paclitaxel; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen I (Experimental): Cisplatin 50 mg/m2 IV Days 1 and 29 plus Volume-directed radiation therapy followed by Carboplatin AUC 5 or 6 plus Paclitaxel 175 mg/m2 q 21 days for 4 cycles
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Regimen II (Active Comparator): Carboplatin AUC 6 plus Paclitaxel 175 mg/m2 q 21 days for 3 cycles followed by Volume-directed radiation therapy followed by Carboplatin AUC 5 or 6 plus Paclitaxel 175 mg/m2 q 21 days for 3 cycles
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Platinol
  Arms: Regimen I
Drug: Carboplatin — Given IV
  Other Names: Paraplatin
Drug: Paclitaxel — Given IV
  Other Names: Taxol
Radiation: Radiation Therapy — Undergo Radiation Therapy
  Other Names: RT; Irradiation

SUMMARY:
To determine if treatment with cisplatin and radiation followed by carbo and taxol reduces the rate of recurrence when compared to sandwich therapy.

DETAILED DESCRIPTION:
To determine if treatment with cisplatin and volume-directed radiation followed by carboplatin and paclitaxel for 4 cycles (experimental arm) reduces the rate of recurrence (increases recurrence-free survival) when compared to sandwich therapy (control arm).

To determine if treatment with cisplatin and volume-directed radiation followed by carboplatin and paclitaxel for 4 cycles (experimental arm) reduces the rate of death (increases survival) when compared to sandwich therapy (control arm).

To compare the regimens with respect to tolerability and acute and late adverse effects of therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Surgical Stage III or IVA endometrial carcinoma per FIGO 2009 staging criteria, including clear cell and serous papillary and undifferentiated carcinomas.
* Surgical Stage III disease includes those patients with positive adnexa, parametrial involvement, tumor invading the serosa, positive pelvic and/or para-aortic nodes, or vaginal involvement.
* Surgical Stage IVA includes patients with bladder or bowel mucosal involvement, but no spread outside the pelvis.
* Patients with FIGO 2009 surgical Stage I or II endometrial clear cell or serous carcinoma and with positive peritoneal cytology.
* Surgery must have included a hysterectomy and bilateral salpingooophorectomy. Pelvic lymph node sampling and para-aortic lymph node sampling are optional.
* Patients with a GOG Performance Status of 0, 1, or 2.
* Patients with adequate organ function, reflected by the following parameters:

WBC ≥ 3000/mcl Absolute neutrophil count (ANC) ≥ 1500/mcl Platelet count ≥ 100,000/mcl SGOT, SGPT, and alkaline phosphatase ≤ 2.5 X upper limit of normal (ULN) Bilirubin ≤ 1.5 X ULN Creatinine ≤ institutional ULN

* Patients must be 18 years of age or older.
* Entry into the study is limited to no more than 8 weeks from the date of surgery.

Exclusion Criteria:

* Patients with carcinosarcoma.
* Patients with recurrent endometrial cancer.
* Patients with residual tumor after surgery (any single site) exceeding 1 cm in maximum dimension.
* Patients who have had pelvic or abdominal radiation therapy.
* Patients with positive pelvic washings as the only extra-uterine disease are NOT eligible if the histology is other than clear cell or papillary serous carcinoma.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of active malignancy within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients with a history of serious co-morbid illness or uncontrolled illnesses that would preclude protocol therapy.
* Patients with an estimated survival of less than three months.
* Patients with FIGO 2009 Stage IVB endometrial cancer.
* Patients with parenchymal liver metastases.
* Patients who have received prior chemotherapy for endometrial cancer.
* Patients with a history of myocardial infarction, unstable angina, or uncontrolled arrhythmia within 3 months from enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | From study entry until disease recurrence, death, or date of last contact, assessed up to 8 years
  RFS will be assessed by radiology tests, patient's clinical symptoms or physical exam.

SECONDARY OUTCOMES:
Overall survival (OS) | from study entry to death or date of last contact, assessed up to 8 years
  OS assessed by the contact with patient in person or by telephone

OTHER OUTCOMES:
Incidence of acute and adverse effects as graded by the NCI Common Toxicity Criteria for Adverse Events version (CTCAE) version 4.0 | From study entry through completion of study treatment, assessed for 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce N Barlin, MD, Principal Investigator — Women's Cancer Care Associates, LLC
Locations (7):
- United States (6):
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Munson Health Care, Traverse City, Michigan
  - Atlantic Health, Morristown, New Jersey
  - Women's Cancer Care Associates, LLC, Albany, New York
  - The Ohio State University, Columbus, Ohio
  - Gunderson Lutheran Medical Foundation, La Crosse, Wisconsin
- CHUM Hopital Notre-Dame, Montreal, Quebec, Canada